CLINICAL TRIAL: NCT00736346
Title: Efficacy of Three Treatment Modalities for Panic Disorder Among Individuals Consulting Emergency Departments for Non Cardiac Chest Pain
Brief Title: Treatment of Panic Disorder Among Individuals Consulting Emergency Departments for Non Cardiac Chest Pain
Acronym: MADONA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Université du Québec a Montréal (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: André Marchand, UQAM
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MOP 81128 (CIHR)
Record Dates: First submitted 2008-08-14; First posted 2008-08-15 (Estimated); Last update posted 2008-08-15 (Estimated); Status verified 2008-08

CONDITIONS: Panic Disorder; Anxiety Disorder; Mental Disorder
Keywords: Panic Disorder; anxiety; chest pain; emergency department; cognitive-behavioral treatment
MeSH Terms: conditions — Panic Disorder; Anxiety Disorders; Mental Disorders; Chest Pain; Emergencies | interventions — Cognitive Behavioral Therapy; Paroxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Active Comparator)
  Interventions: Behavioral: Brief cognitive-behavioral treatment for Panic Disorder
- 2 (Active Comparator)
  Interventions: Behavioral: Cognitive-Behavior Therapy for Panic Disorder
- 3 (Active Comparator)
  Interventions: Drug: paroxetine
- 4 (No Intervention)

INTERVENTIONS:
Behavioral: Brief cognitive-behavioral treatment for Panic Disorder — One two-hour session of cognitive-behavior therapy for panic disorder
  Arms: 1
Behavioral: Cognitive-Behavior Therapy for Panic Disorder — Seven one-hour sessions of cognitive-behavior therapy for panic disorder
  Arms: 2
Drug: paroxetine — 40 mg die, for 6 months
  Arms: 3

SUMMARY:
The purpose of this study is to assess the impact of three different treatment modalities on panic symptoms, quality of life and use of health services among individuals consulting an emergency department for non cardiac chest pain and having Panic Disorder.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 and over
* Mastered oral and written French
* Consulted an emergency department for chest pain with very low risk of coronary disease (normal ECG and blood tests)
* Met criteria for Panic Disorder

Exclusion Criteria:

* Chest pain with an obvious medical origin (obvious trauma or abnormal pulmonary x-rays)
* Had received cognitive-behavior therapy for Panic Disorder in the last six months
* Cognitive impairment preventing the completion of psychological assessment
* Past or present psychotic episode, Bipolar Disorder, or organic mental disorder
* Current Abuse or Dependence Disorder
* If another Mental Disorder is present, its severity was equal or inferior to the severity of Panic Disorder
* Current medical condition preventing the participant from receiving pharmacological of cognitive-behavior treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2005-10; Primary Completion 2009-12 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
Panic Disorder diagnosis | Pre and posttreatment, and 3, 6 and 12 months after treament

SECONDARY OUTCOMES:
Panic symptomatology, psychological distress, quality of life, and use of health services | Pre and posttreatment, and 3, 6 and 12 months after treatment

CONTACTS AND LOCATIONS:
Overall Officials: André Marchand, PhD, Principal Investigator — Université du Québec a Montréal
Locations (3):
- Canada (3):
  - Hôtel-Dieu de Lévis, Lévis, Quebec
  - Institut de Cardiologie de Montréal (Montreal Heart Institute), Montreal, Quebec
  - Hôpital du Sacré-Coeur de Montréal, Montreal, Quebec

REFERENCES:
- [Derived] Foldes-Busque G, Hamel S, Belleville G, Fleet R, Poitras J, Chauny JM, Vadeboncoeur A, Lavoie KL, Marchand A. Factors associated with pain level in non-cardiac chest pain patients with comorbid panic disorder. Biopsychosoc Med. 2016 Oct 18;10:30. doi: 10.1186/s13030-016-0081-5. eCollection 2016. PMID 27777612